CLINICAL TRIAL: NCT06002269
Title: A Home-based Lifestyle Intervention for Optimizing Surgical Outcomes Among Urinary Bladder Cancer Patients: the BOOST Study
Brief Title: A Home-based Lifestyle Intervention for Optimizing Surgical Outcomes Among Urinary Bladder Cancer Patients
Acronym: BOOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCI150155
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Cystectomy; Chemotherapy
Keywords: Surgery; Weight Loss; Urinary; Lifestyle; Cystectomy; Malnutrition; Chemotherapy; Diet; Exercise
MeSH Terms: conditions — Urinary Bladder Neoplasms; Weight Loss; Malnutrition; Motor Activity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: BOOST Box intervention compared with usual care.
Who Masked: Care Provider
Masking Description: Dietitians will be masked to study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOOST Box Intervention (Experimental): Baseline: Questionnaires (FACT-Bl-Cys, mPG-SGA, Short 2012, FAACT, Godin, TCC), exercise prescription, compensation.
  Pre-Surgery: Dietitian consultation, at least 3-weeks and up to 6-weeks of Boost Box deliveries and check-ins (nutritional intervention), up to 6 weeks of exercise intervention and logs, ASA Food Record (x2), compensation Post-Surgery: post-surgery surveys once (FACT-Bl-Cys, mPG-SGA, FAACT, Godin), 6 weeks of Boost Box deliveries and check-ins (nutritional intervention), 6 weeks of exercise intervention and logs, weekly hunger check-in, ASA Food Record (x2), Dietitian consultation, compensation.
  Follow-up (estimated 6 months after baseline) : 6-month questionnaire, compensation.
  Compensation total: up to $100 via electronic gift card.
  Interventions: Combination Product: Dietary and Exercise Intervention
- Usual Care (No Intervention): Baseline: Questionnaires (FACT-Bl-Cys, mPG-SGA, Short 2012, FAACT, Godin, TCC), compensation.
  Pre-Surgery: Dietitian consultation, ASA Food Record (x2), compensation. Post-Surgery: post-surgery surveys once (FACT-Bl-Cys, mPG-SGA, FAACT, Godin), Dietitian consultation, ASA Food Record (x2), compensation.
  Follow-up (estimated 6 months after baseline): 6-month questionnaire, compensation.
  Compensation total: up to $100 via electronic gift card.

INTERVENTIONS:
Combination Product: Dietary and Exercise Intervention — Participants will receive food ingredients and recipes to be made and consumed for each meal, every day for a period of 3-6 weeks before surgery and 6-weeks after surgery. The menu is designed as a high protein, high calorie diet meeting targets for omega-3 fatty acids, vitamin A, and arginine (immunonutrition meal plan). In addition, participants will receive an individualized exercise prescription to be performed at home using theraband resistance bands.
  Arms: BOOST Box Intervention

SUMMARY:
The purpose of this study is to test a randomized, controlled diet and physical activity intervention designed to be simple and address barriers to participation in lifestyle intervention among 16 urinary bladder cancer patients.

Aim 1 is to test the feasibility and acceptability of a novel, peri-operative lifestyle intervention, "The Boost Box", among bladder cancer patients receiving cystectomy with or without neo-adjuvant chemotherapy.

Aim 2 is to measure the feasibility of collecting data on the intervention effects on complication rate, nutritional status, weight loss, and quality of life post-surgery among bladder cancer patients receiving cystectomy ± neoadjuvant therapy. Secondarily, we will determine the magnitude of association between study group and outcomes to inform power calculations in a future, well-powered trial.

Participants will:

* attend two dietetic consultations at baseline and post-surgical recovery where nutritional status will be evaluated with patient-generated subjective global assessment (PG-SGA)
* complete baseline questionnaires (TCC, FACT-BI-Cys, Short 2012, FAACT, Godin)
* receive weekly BOOST boxes
* complete pre-surgery weekly BOOST check ins
* complete post-surgery weekly BOOST check ins
* complete an ASA food recall pre and post-surgery
* complete an exercise familiarization consult
* record weekly resistance and aerobic exercise performed at home
* complete a 6 month follow-up questionnaire
* receive compensation

Researchers will compare to a Usual Care group to determine differences that could be attributed to the BOOST Box intervention.

DETAILED DESCRIPTION:
Urinary bladder cancer is the fourth leading cancer in men in the US, leading to 18,000 deaths among men and women annually.1 The survival rate is 69% for localized disease, 36% for regional disease, and only 5% for metastatic disease.2 Bladder cancer patients often present with non-muscle invasive bladder cancer (NMIBC) and are treated with chemotherapy or immunotherapy delivered locally in the bladder. Patients with muscle- invasive bladder cancer or intravesical therapy-refractory disease undergo cystectomy. Weight loss, frailty, sarcopenia, and malnutrition are commonplace among urinary bladder cancer patients, all being associated with treatment-related complications including susceptibility to infection, poor prognosis and quality of life.3 Medical nutrition therapy is indicated in this population that generally has poor diet quality4-7 to achieve or maintain a healthy body weight, preserve lean body mass, minimize nutrition-related side effects, and maximize quality of life.8-10 Yet, only a handful of dietary interventions have been conducted among urinary bladder cancer patients, and no studies of diet intervention coupled with exercise prescription, with the goal of improving treatment outcomes in this population. Pre- and postoperative nutrition support has been linked to reduced hospital length of stay,11 and lower postoperative complications like infection. Immunonutrition interventions, which comprise of supplements or food/drinks high in vitamin A, fish oil or omega-3 fatty acids, and specific amino acids like arginine, have also been shown to lower postoperative complications in cystectomy patients and other cancer populations.12-15 In patients receiving chemotherapy or radiation, immunonutrition also appears to reduce mucositis and weight loss.16 Furthermore, resistance exercise promotes maintenance or increase in muscle mass, particularly among individuals with sarcopenia.17

Little is known about the trajectory of dietary intake after bladder cancer diagnosis, and the specific nutritional needs of this population in diverse settings where health disparities exist, such as among rural or socio- economically disadvantaged patients.18 There is also a critical need to develop and test interventions that are simple, scalable, durable, and cost-effective,4, 19 and that address food insecurity.20 Given these major research gaps, we will implement a novel, peri-operative lifestyle intervention rooted in Social Cognitive Theory (SCT)21, 22 that uses food/ingredient, menu and recipe provision coupled with resistance exercise recommendations and tools provided in the "Boost Box", mailed to participants over 12-weeks. The intervention builds self-efficacy and behavioral capability in preparing meals to support nutrition goals and addresses social determinants of health in underserved populations by tackling food insecurity.23 Community partnerships will build the foundation for scaling up lifestyle intervention for cancer patients in Utah. Expanding the availability of evidence-based options for nutrition and physical activity counseling for cancer patients and survivors has been identified as a major need.24 Our proposed study is multidisciplinary and community-focused by partnering with the University of Utah Center for Community Nutrition and their established partners (e.g., Waste Less Solutions, Wasatch Community Gardens, Food Recovery Network, Utah Food Bank, Dairy West, and commercial grocers like Smiths and Harmons) to roll out the intervention in the community. Indeed, community and home-based lifestyle interventions improve physical functioning and clinical outcomes among cancer survivors and are cost-effective.25, 26 Delivering diet and physical activity education using a home-based 'Blue Apron' type approach in partnership with the community is highly novel.

Urinary bladder cancer is the fourth leading cancer in men in the US and accounts for over 18,000 deaths among both men and women annually.1 About three quarters of bladder cancer patients present with non- muscle invasive bladder cancer and are treated with chemotherapy or immunotherapy delivered locally in the bladder, or cystectomy alone in intravesical-refractory or extensive disease. Muscle-invasive bladder cancer treatment includes neoadjuvant cisplatin-based chemotherapy followed by radical cystectomy. Cisplatin- ineligible patients proceed with cystectomy and those who are too sick or frail for cystectomy receive chemotherapy followed by local radiation. Weight loss is a common occurrence post-radical cystectomy, and is associated with malnutrition3 and poor overall survival.34 Moreover, up to 70% of bladder cancer patients, particularly those with frailty, present with sarcopenia, a condition of reduced skeletal muscle mass and function that is an independent poor prognostic factor35 linked to medical complications and quality of life.36 In all, this population has a 60% complication rate by 90-days,37 from urinary tract infections to bowel obstruction.

Nutrition is a vital component of chemotherapy tolerability and preparation for and recovery after cystectomy38 to prevent or resolve nutrient deficiencies, achieve or maintain a healthy body weight, preserve lean body mass, minimize nutrition-related side effects, and maximize quality of life.4, 8-10, 39 Diet quality is generally poor among adult cancer survivors in the United States.4 Bladder cancer is especially prevalent in developed countries with Western style dietary patterns and high levels of obesity,2, 40 with significant socioeconomic and geographic disparities observed.18, 41 Indeed, rural compared with urban residence is associated with elevated cancer-specific and other cause mortality among bladder cancer survivors.41 In addition, improvement in diet quality among cancer survivors undergoing dietary intervention has been found to be smaller in rural than urban patients. Yet, despite the biologically plausible role of diet in the etiology of bladder cancer, and the potent effects of treatment on nutritional status and weight loss in this population, remarkably few studies have evaluated either pre- or post-diagnosis diet in association with outcomes after bladder cancer diagnosis, nor implemented dietary intervention among bladder cancer patients to optimize their treatment outcomes.42

We will address this immense research gap by testing a randomized, controlled diet and physical activity trial designed to address barriers to participation in lifestyle intervention among 16 urinary bladder cancer patients (50% rural; 50% no college education). Baseline and post-surgical recovery nutritional status will be evaluated with patient-generated subjective global assessment (PG-SGA).43, 44 Diet will be assessed with 3-day food record during the first 6-months post-diagnosis. In the intervention arm, patients will be mailed a "Boost Box" weekly for 6-weeks before and 6-weeks after surgery, prepared by our community partners, containing food ingredients. We will work with the University of Utah Center for Community Nutrition to mail curriculum boxes with a menu and recipes for a high protein, immunonutrition-tailored diet (i.e., arginine, vitamin A, and omega-3 rich foods/beverages), and resistance bands (Theraband) with strength training guidelines.3,

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years or older.
2. Newly diagnosed urinary bladder cancer patients indicated for cystectomy with or without neo-adjuvant therapy; Treated with surgery at the Huntsman Cancer Institute
3. Have reliable, consistence access to the internet for study procedures

Inclusion of Individuals across the Lifespan: The proposed trial will enroll 20 adults who have been diagnosed with bladder cancer. The age range of participants to be recruited is 18 years or older. Bladder cancer is generally a disease of older age and is exceedingly rare in children. According to the American Cancer Society, average age at diagnosis is 73.1 Therefore, we are unable to include children in this trial.

Inclusion of Women, Minorities, and Children: It is anticipated that 20% will be female; 80% male. Racial distribution is projected to be as follows: 97% white, 1% Native Hawaiian or Pacific Islander; 1% American Indian/ Alaska Native; 1% Asian; <1% Black. Approximately 96% will be Non-Hispanic.

Exclusion Criteria:

1. Special dietary requirements (i.e., allergies and intolerances, or other clinically prescribed diet).
2. Unable to provide informed consent or read, write, or fill in questionnaires in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of BOOST Box Intervention | From enrollment to the 6-month follow-up survey
  Feasibility of a novel, peri-operative lifestyle intervention, "The Boost Box", among bladder cancer patients receiving cystectomy with or without neo-adjuvant chemotherapy.
  Feasibility metrics include: % consented/referred; attrition as a function of time; % questionnaires completed; % meals prepared and consumed. Feasibility criteria: >70% patients consented and retained; completed all questionnaires; prepared/consumed Boost Box meals ≥5/7 days/week; and adhered to resistance band exercise ≥2 days/week. Fidelity criteria: 90% protocol checklist items delivered as intended.
Acceptability of BOOST Box Intervention | From enrollment to the 6-month follow-up survey
  Acceptability of a novel, peri-operative lifestyle intervention, "The Boost Box", among bladder cancer patients receiving cystectomy with or without neo-adjuvant chemotherapy.
  Acceptability of the intervention delivery and menus/recipes will be evaluated by administering an anonymous questionnaire incorporating both Likert scale questions and space for open-ended responses.

SECONDARY OUTCOMES:
Malnutrition assessment | mPG-SGA, FAACT, and Short 2012 at baseline and then mPG-SGA and FAACT again six weeks post-surgery. ASA24 during six weeks pre and post-surgery
  Surveys and Questionnaires used will be the Modified Patient-Generated Subjective Global Assessment (mPG-SGA), Functional Assessment of Anorexia and Cachexia Therapy (FAACT), U.S.Household Food Security Survey Module: Six Item Short Form (Short 2012), and Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) food consumption log to calculate a Healthy Eating Index (HEI) which will define diet quality (a higher score indicates a healthier diet).
Surgical complication rate | 30 and 60 days post-surgery
  The following information is to be abstracted from medical charts: 30- and 90-day post-surgery complication rates including wound infections; Urinary Tract Infection (UTI); infectious complications; blood clots; readmissions; failure to thrive; dehydration; re-operations.
Body weight | From enrollment to the 6-month follow-up survey
  Participant weight measurements will be collected through participant self-reporting using a digital scale provided by the study and through medical record abstraction.
Quality of Life (Physical, social, emotional, functional well-being, and a bladder cancer subscale) | FACT-BI-Cys used from baseline to the 6-month follow-up survey
  Questionnaire used will be the Functional Assessment of Cancer Therapy - Bladder - Cystectomy (FACT-Bl-Cys).

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Playdon, PhD, MPH, Principal Investigator — University of Utah NUIP Department and Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Tobert CM, Hamilton-Reeves JM, Norian LA, Hung C, Brooks NA, Holzbeierlein JM, Downs TM, Robertson DP, Grossman R, Nepple KG. Emerging Impact of Malnutrition on Surgical Patients: Literature Review and Potential Implications for Cystectomy in Bladder Cancer. J Urol. 2017 Sep;198(3):511-519. doi: 10.1016/j.juro.2017.01.087. Epub 2017 Mar 9. PMID 28286066
- [Background] Gregg JR, Cookson MS, Phillips S, Salem S, Chang SS, Clark PE, Davis R, Stimson CJ Jr, Aghazadeh M, Smith JA Jr, Barocas DA. Effect of preoperative nutritional deficiency on mortality after radical cystectomy for bladder cancer. J Urol. 2011 Jan;185(1):90-6. doi: 10.1016/j.juro.2010.09.021. Epub 2010 Nov 12. PMID 21074802
- [Background] Hansen TTD, Omland LH, von Heymann A, Johansen C, Clausen MB, Suetta C, Pappot H, Rafn BS. Development of Sarcopenia in Patients With Bladder Cancer: A Systematic Review. Semin Oncol Nurs. 2021 Feb;37(1):151108. doi: 10.1016/j.soncn.2020.151108. Epub 2021 Jan 8. PMID 33431235
- [Background] Grimberg DC, Shah A, Molinger J, Whittle J, Gupta RT, Wischmeyer PE, McDonald SR, Inman BA. Assessments of frailty in bladder cancer. Urol Oncol. 2020 Sep;38(9):698-705. doi: 10.1016/j.urolonc.2020.04.036. Epub 2020 May 22. PMID 32451229
- [Background] Maibom SL, Joensen UN, Poulsen AM, Kehlet H, Brasso K, Roder MA. Short-term morbidity and mortality following radical cystectomy: a systematic review. BMJ Open. 2021 Apr 14;11(4):e043266. doi: 10.1136/bmjopen-2020-043266. PMID 33853799
- [Background] Jensen BT, Lauridsen SV, Jensen JB. Optimal Delivery of Follow-Up Care After Radical Cystectomy for Bladder Cancer. Res Rep Urol. 2020 Oct 14;12:471-486. doi: 10.2147/RRU.S270240. eCollection 2020. PMID 33117747
- [Background] Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz AL, Bandera EV, Hamilton KK, Grant B, McCullough M, Byers T, Gansler T. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012 Jul-Aug;62(4):243-74. doi: 10.3322/caac.21142. Epub 2012 Apr 26. PMID 22539238
- [Background] Prado CM, Purcell SA, Laviano A. Nutrition interventions to treat low muscle mass in cancer. J Cachexia Sarcopenia Muscle. 2020 Apr;11(2):366-380. doi: 10.1002/jcsm.12525. Epub 2020 Jan 8. PMID 31916411
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] Keaver L, Houlihan C, O'Callaghan N, LaVertu AE, Ding X, Zhang FF. Evidence-based nutrition guidelines for cancer survivors in Europe: a call for action. Eur J Clin Nutr. 2022 Jun;76(6):819-826. doi: 10.1038/s41430-021-01036-8. Epub 2021 Oct 29. PMID 34716363
- [Background] Demark-Wahnefried W, Rogers LQ, Alfano CM, Thomson CA, Courneya KS, Meyerhardt JA, Stout NL, Kvale E, Ganzer H, Ligibel JA. Practical clinical interventions for diet, physical activity, and weight control in cancer survivors. CA Cancer J Clin. 2015 May-Jun;65(3):167-89. doi: 10.3322/caac.21265. Epub 2015 Feb 13. PMID 25683894
- [Background] Saginala K, Barsouk A, Aluru JS, Rawla P, Padala SA, Barsouk A. Epidemiology of Bladder Cancer. Med Sci (Basel). 2020 Mar 13;8(1):15. doi: 10.3390/medsci8010015. PMID 32183076
- [Background] Jochems SHJ, Van Osch FHM, Bryan RT, Wesselius A, van Schooten FJ, Cheng KK, Zeegers MP. Impact of dietary patterns and the main food groups on mortality and recurrence in cancer survivors: a systematic review of current epidemiological literature. BMJ Open. 2018 Feb 19;8(2):e014530. doi: 10.1136/bmjopen-2016-014530. PMID 29459359
- [Background] Lee E, Zhu J, Velazquez J, Bernardo R, Garcia J, Rovito M, Hines RB. Evaluation of Diet Quality Among American Adult Cancer Survivors: Results From 2005-2016 National Health and Nutrition Examination Survey. J Acad Nutr Diet. 2021 Feb;121(2):217-232. doi: 10.1016/j.jand.2020.08.086. Epub 2020 Nov 3. PMID 33158797
- [Background] Deuker M, Stolzenbach LF, Colla Ruvolo C, Nocera L, Tian Z, Roos FC, Becker A, Kluth LA, Tilki D, Shariat SF, Saad F, Chun FKH, Karakiewicz PI. Bladder cancer stage and mortality: urban vs. rural residency. Cancer Causes Control. 2021 Feb;32(2):139-145. doi: 10.1007/s10552-020-01366-1. Epub 2020 Nov 23. PMID 33230694
- [Background] Oberle AD, West JM, Tobert CM, Conley GL, Nepple KG. Optimizing Nutrition Prior to Radical Cystectomy. Curr Urol Rep. 2018 Oct 18;19(12):99. doi: 10.1007/s11934-018-0854-4. PMID 30338466
- [Background] Cunha Cde M, Sampaio Ede J, Varjao ML, Factum CS, Ramos LB, Barreto-Medeiros JM. Nutritional assessment in surgical oncology patients: a comparative analysis between methods. Nutr Hosp. 2014 Nov 1;31(2):916-21. doi: 10.3305/nh.2015.31.2.7715. PMID 25617581
- [Background] Bauer J, Capra S, Ferguson M. Use of the scored Patient-Generated Subjective Global Assessment (PG-SGA) as a nutrition assessment tool in patients with cancer. Eur J Clin Nutr. 2002 Aug;56(8):779-85. doi: 10.1038/sj.ejcn.1601412. PMID 12122555
- [Background] Hamilton-Reeves JM, Stanley A, Bechtel MD, Yankee TM, Chalise P, Hand LK, Lee EK, Smelser W, Mirza M, Wyre H, Hull H, Carlson SE, Holzbeierlein JM. Perioperative Immunonutrition Modulates Inflammatory Response after Radical Cystectomy: Results of a Pilot Randomized Controlled Clinical Trial. J Urol. 2018 Aug;200(2):292-301. doi: 10.1016/j.juro.2018.03.001. Epub 2018 Mar 6. PMID 29518432
- [Background] Hamilton-Reeves JM, Bechtel MD, Hand LK, Schleper A, Yankee TM, Chalise P, Lee EK, Mirza M, Wyre H, Griffin J, Holzbeierlein JM. Effects of Immunonutrition for Cystectomy on Immune Response and Infection Rates: A Pilot Randomized Controlled Clinical Trial. Eur Urol. 2016 Mar;69(3):389-92. doi: 10.1016/j.eururo.2015.11.019. Epub 2015 Nov 30. PMID 26654125
- [Background] Solerte SB, Gazzaruso C, Bonacasa R, Rondanelli M, Zamboni M, Basso C, Locatelli E, Schifino N, Giustina A, Fioravanti M. Nutritional supplements with oral amino acid mixtures increases whole-body lean mass and insulin sensitivity in elderly subjects with sarcopenia. Am J Cardiol. 2008 Jun 2;101(11A):69E-77E. doi: 10.1016/j.amjcard.2008.03.004. PMID 18514630
- [Background] Gopalakrishna A, Chang A, Longo TA, Fantony JJ, Harrison MR, Wischmeyer PE, Inman BA. Dietary patterns and health-related quality of life in bladder cancer survivors. Urol Oncol. 2018 Oct;36(10):469.e21-469.e29. doi: 10.1016/j.urolonc.2018.06.001. Epub 2018 Aug 17. PMID 30126776
- [Background] Westhoff E, Wu X, Kiemeney LA, Lerner SP, Ye Y, Huang M, Dinney CP, Vrieling A, Tu H. Dietary patterns and risk of recurrence and progression in non-muscle-invasive bladder cancer. Int J Cancer. 2018 May 1;142(9):1797-1804. doi: 10.1002/ijc.31214. Epub 2017 Dec 26. PMID 29235103
- [Background] Westhoff E, Witjes JA, Fleshner NE, Lerner SP, Shariat SF, Steineck G, Kampman E, Kiemeney LA, Vrieling A. Body Mass Index, Diet-Related Factors, and Bladder Cancer Prognosis: A Systematic Review and Meta-Analysis. Bladder Cancer. 2018 Jan 20;4(1):91-112. doi: 10.3233/BLC-170147. PMID 29430510
- [Background] Declercq P, De Win G, Van der Aa F, Beels E, Van der Linden L, Van Poppel H, Willems L, Spriet I. Reduced length of stay in radical cystectomy patients with oral versus parenteral post-operative nutrition protocol. Int J Clin Pharm. 2015 Apr;37(2):379-86. doi: 10.1007/s11096-015-0072-9. Epub 2015 Feb 10. PMID 25666940
- [Background] Bertrand J, Siegler N, Murez T, Poinas G, Segui B, Ayuso D, Gres P, Wagner L, Thuret R, Costa P, Droupy S. Impact of preoperative immunonutrition on morbidity following cystectomy for bladder cancer: a case-control pilot study. World J Urol. 2014 Feb;32(1):233-7. doi: 10.1007/s00345-013-1229-6. Epub 2013 Dec 21. PMID 24362882
- [Background] Kanekiyo S, Takeda S, Iida M, Nishiyama M, Kitahara M, Shindo Y, Tokumitsu Y, Tomochika S, Tsunedomi R, Suzuki N, Abe T, Yoshino S, Hazama S, Ueno T, Nagano H. Efficacy of perioperative immunonutrition in esophageal cancer patients undergoing esophagectomy. Nutrition. 2019 Mar;59:96-102. doi: 10.1016/j.nut.2018.08.006. Epub 2018 Aug 22. PMID 30468936
- [Background] Yu K, Zheng X, Wang G, Liu M, Li Y, Yu P, Yang M, Guo N, Ma X, Bu Y, Peng Y, Han C, Yu K, Wang C. Immunonutrition vs Standard Nutrition for Cancer Patients: A Systematic Review and Meta-Analysis (Part 1). JPEN J Parenter Enteral Nutr. 2020 Jul;44(5):742-767. doi: 10.1002/jpen.1736. Epub 2019 Nov 11. PMID 31709584
- [Background] Buzquurz F, Bojesen RD, Grube C, Madsen MT, Gogenur I. Impact of oral preoperative and perioperative immunonutrition on postoperative infection and mortality in patients undergoing cancer surgery: systematic review and meta-analysis with trial sequential analysis. BJS Open. 2020 Oct;4(5):764-775. doi: 10.1002/bjs5.50314. Epub 2020 Jun 23. PMID 32573977
- [Background] Zheng X, Yu K, Wang G, Liu M, Li Y, Yu P, Yang M, Guo N, Ma X, Bu Y, Peng Y, Han C, Yu K, Wang C. Effects of Immunonutrition on Chemoradiotherapy Patients: A Systematic Review and Meta-Analysis. JPEN J Parenter Enteral Nutr. 2020 Jul;44(5):768-778. doi: 10.1002/jpen.1735. Epub 2019 Nov 11. PMID 31709589
- [Background] Jang MK, Park C, Tussing-Humphreys L, Fernhall B, Phillips S, Doorenbos AZ. The Effectiveness of Sarcopenia Interventions for Cancer Patients Receiving Chemotherapy: A Systematic Review and Meta-analysis. Cancer Nurs. 2023 Mar-Apr 01;46(2):E81-E90. doi: 10.1097/NCC.0000000000000957. PMID 34054070
- [Background] Jones LW, Courneya KS, Fairey AS, Mackey JR. Effects of an oncologist's recommendation to exercise on self-reported exercise behavior in newly diagnosed breast cancer survivors: a single-blind, randomized controlled trial. Ann Behav Med. 2004 Oct;28(2):105-13. doi: 10.1207/s15324796abm2802_5. PMID 15454357
- [Background] Feathers A, Aycinena AC, Lovasi GS, Rundle A, Gaffney AO, Richardson J, Hershman D, Koch P, Contento I, Greenlee H. Food environments are relevant to recruitment and adherence in dietary modification trials. Nutr Res. 2015 Jun;35(6):480-8. doi: 10.1016/j.nutres.2015.04.007. Epub 2015 Apr 16. PMID 25981966
- [Background] Sremanakova J, Sowerbutts AM, Todd C, Cooke R, Burden S. Systematic Review of Behaviour Change Theories Implementation in Dietary Interventions for People Who Have Survived Cancer. Nutrients. 2021 Feb 13;13(2):612. doi: 10.3390/nu13020612. PMID 33668596
- [Background] Trego ML, Baba ZM, DiSantis KI, Longacre ML. Food insecurity among adult cancer survivors in the United States. J Cancer Surviv. 2019 Aug;13(4):641-652. doi: 10.1007/s11764-019-00783-9. Epub 2019 Jul 11. PMID 31297721
- [Background] Basen-Engquist K, Alfano CM, Maitin-Shepard M, Thomson CA, Schmitz KH, Pinto BM, Stein K, Zucker DS, Syrjala KL, Fallon E, Doyle C, Demark-Wahnefried W. Agenda for Translating Physical Activity, Nutrition, and Weight Management Interventions for Cancer Survivors into Clinical and Community Practice. Obesity (Silver Spring). 2017 Nov;25 Suppl 2(Suppl 2):S9-S22. doi: 10.1002/oby.22031. PMID 29086526
- [Background] Swartz MC, Lewis ZH, Lyons EJ, Jennings K, Middleton A, Deer RR, Arnold D, Dresser K, Ottenbacher KJ, Goodwin JS. Effect of Home- and Community-Based Physical Activity Interventions on Physical Function Among Cancer Survivors: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2017 Aug;98(8):1652-1665. doi: 10.1016/j.apmr.2017.03.017. Epub 2017 Apr 17. PMID 28427925
- [Background] Demark-Wahnefried W, Morey MC, Sloane R, Snyder DC, Miller PE, Hartman TJ, Cohen HJ. Reach out to enhance wellness home-based diet-exercise intervention promotes reproducible and sustainable long-term improvements in health behaviors, body weight, and physical functioning in older, overweight/obese cancer survivors. J Clin Oncol. 2012 Jul 1;30(19):2354-61. doi: 10.1200/JCO.2011.40.0895. Epub 2012 May 21. PMID 22614994
- [Background] De Groot LM, Lee G, Ackerie A, van der Meij BS. Malnutrition Screening and Assessment in the Cancer Care Ambulatory Setting: Mortality Predictability and Validity of the Patient-Generated Subjective Global Assessment Short form (PG-SGA SF) and the GLIM Criteria. Nutrients. 2020 Jul 30;12(8):2287. doi: 10.3390/nu12082287. PMID 32751724
- [Background] Arends J, Baracos V, Bertz H, Bozzetti F, Calder PC, Deutz NEP, Erickson N, Laviano A, Lisanti MP, Lobo DN, McMillan DC, Muscaritoli M, Ockenga J, Pirlich M, Strasser F, de van der Schueren M, Van Gossum A, Vaupel P, Weimann A. ESPEN expert group recommendations for action against cancer-related malnutrition. Clin Nutr. 2017 Oct;36(5):1187-1196. doi: 10.1016/j.clnu.2017.06.017. Epub 2017 Jun 23. PMID 28689670
- [Background] Krebs-Smith SM, Pannucci TE, Subar AF, Kirkpatrick SI, Lerman JL, Tooze JA, Wilson MM, Reedy J. Update of the Healthy Eating Index: HEI-2015. J Acad Nutr Diet. 2018 Sep;118(9):1591-1602. doi: 10.1016/j.jand.2018.05.021. PMID 30146071